CLINICAL TRIAL: NCT00963261
Title: Side-effect Management for Patients With Malignant Melanoma Undergoing Treatment With Interferon Alpha (IFN-α)- Diagnosis and Therapy -
Brief Title: Quality of Life and Psychological Well-being in Patients With Malignant Melanoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Freiburg (Other)
Collaborators: Essex Pharma GmbH (Industry); Universitätsklinikum Köln (Other)
Responsible Party: Katrin Reuter, PhD; Dorothee Nashan, MD, University Medical Center Freiburg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PO5098
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2010-06

CONDITIONS: Malignant Melanoma
Keywords: melanoma; interferon-a; quality of life; psychological distress; depressive symptoms; side effects
MeSH Terms: conditions — Melanoma; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- psycho-oncological intervention (Experimental): stepped care psycho-oncological intervention
  Interventions: Behavioral: psycho-oncological intervention
- control group (No Intervention)

INTERVENTIONS:
Behavioral: psycho-oncological intervention — stepped care treatment program with different elements (patient information, exercise, psychoeducation, individual and group therapy, psycho-pharmacology)
  Arms: psycho-oncological intervention

SUMMARY:
The purpose of this study is to analyse the physical and psychological side-effects in the course of treatment with IFN-alpha. The effectiveness of a specific intervention for the management of these side-effects is evaluated.

DETAILED DESCRIPTION:
Today, the consideration of the side effects of intensive treatment measures and their influence on quality of life are regarded as standard procedures in oncology. Quality of life measurements have found their way into clinical studies as patient-reported outcomes. In comparison to other tumor types, the field of dermato-oncology has had less research activity concerning quality of life. However, in recent years more attention has been paid to health related quality of life in malignant melanoma patients, especially under adjuvant treatment with interferon-alpha. Data about high dose IFN-α treatment, especially from the USA, show that there are significant physical and psychological side effects, such as fatigue and depression, which often lead to dosage reduction or termination of treatment. As yet, there are very few systematic studies about low dose IFN-α treatment, especially in regard to the side effects during the course of the disease.

Concerning treatment side-effects it is known throughout various areas of oncology that specific psycho-oncological interventions assist in the patients' adaptation to the illness and handling of the side effects of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Documented and proven stage Ib up to stage IIIc malignant melanoma
* No clinical and radiological evidence or suspicion of persistent disease
* Treatment with IFN-α within a study or analog treatment schedule with IFN-α
* ECOG performance status < 2
* Constant after care
* Informed consent to participate in the study
* melanoma diagnosis within the last 5 years or therapy, recurrence or progression within this period of time.

Exclusion Criteria:

* Inoperable lymph nodes- or distant metastases
* Tumors of other origins or localisations within the past 10 years
* Severe and permanent infectious diseases, e. g. HIV or hepatitis
* Participation in other treatment studies apart from IFN-α
* Insufficient knowledge of German language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-02 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Changes in quality of life | 1 year

SECONDARY OUTCOMES:
Changes in fatigue | 1 year
Changes in psychological distress | 1 year
Changes in depressive syndrome | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Reuter, PhD, Principal Investigator — University Medical Center Freiburg, Department of Psychiatry and Psychotherapy; Dorothee Nashan, MD, Principal Investigator — University Medical Center, Department of Dermatology
Locations (2):
- Germany (2):
  - University Medical Center Collogne, Department of Dermatology, Cologne
  - University Medical Center Freiburg, Department of Dermatology, Freiburg im Breisgau

REFERENCES:
- [Derived] Reuter K, Albrecht K, Seelig H, Meiss F, Mauch C, Kreuzberg N, Nashan D. Health-related quality of life, fatigue, and depression under low-dose IFN-alpha therapy in melanoma patients. J Immunother. 2014 Nov-Dec;37(9):461-7. doi: 10.1097/CJI.0000000000000057. PMID 25304729
- [Derived] Albrecht KJ, Nashan D, Meiss F, Bengel J, Reuter K. Shared decision making in dermato-oncology: preference for involvement of melanoma patients. Melanoma Res. 2014 Feb;24(1):68-74. doi: 10.1097/CMR.0000000000000030. PMID 24136099
- [Derived] Albrecht K, Droll H, Giesler JM, Nashan D, Meiss F, Reuter K. Self-efficacy for coping with cancer in melanoma patients: its association with physical fatigue and depression. Psychooncology. 2013 Sep;22(9):1972-8. doi: 10.1002/pon.3238. Epub 2013 Jan 3. PMID 23288588